CLINICAL TRIAL: NCT00762931
Title: Neurostimulation for the Relief of Acute Bronchoconstriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-01
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: bronchoconstriction; neuromodulation; neurostimulation; vagus nerve stimulation; vagal nerve stimulation; nVNS; VNS; non invasive; gammacore
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resolve Stimulator and Proximity Lead (Experimental): An electrical neurostimulation signal will be applied to the neck via subcutaneous lead placement for vagal nerve stimulation, all subjects will receive active treatment
  Interventions: Device: Resolve Stimulator and Proximity Lead

INTERVENTIONS:
Device: Resolve Stimulator and Proximity Lead — An electrical neurostimulation signal will be applied to the neck via subcutaneous lead placement for vagal nerve stimulation

SUMMARY:
The goal of this study is to validate design for the Resolve™ Stimulator and Proximity Electrode and the associated procedure to quickly and safely place an electrode into the neck, in the vicinity of the vagus nerve by a physician in either the Emergency Department or other appropriate hospital inpatient setting (e.g., ICU). The secondary goal is to confirm that the electrical signal being delivered via this electrode rapidly counters bronchoconstriction and improves airway flow.

DETAILED DESCRIPTION:
The present study is to evaluate the safety of a new neurostimulator device, the Resolve Stimulator and Proximity Lead™, which comprises an external electrical signal generator coupled to temporary electrode that is percutaneously inserted in the neck.

Sponsor believes, based on animal testing data provided as well as consultations with physicians who regularly treat patients suffering from attacks of acute bronchoconstriction in ER and inpatient hospital settings, that this device could be used in the skilled care hospital setting to help rapidly relax the smooth muscle in the airway, relieving a clinically significant portion of the bronchoconstriction suffered by patients experiencing moderate to severe asthma attacks, allowing more effective delivery of inhaled medications to restore the patient to his or her baseline respiration status.

ELIGIBILITY:
Inclusion Criteria:

* Male / Female, Age 18-65
* Subject declares a medical history of asthma or sufficient prior clinical experience/records exists to confirm the subject has received a diagnosis of bronchoconstriction
* Completed >1 hrs of conventional breathing and related medication treatments without improvement in FEV1 to > 70% predicted
* Able to give Informed Consent

Exclusion Criteria:

* Scaring / abscess other problems with neck at electrode placement site
* Known or suspected carotid artery disease (i.e. bruits or history of stenosis)
* Suspected or confirmed coagulopathy
* Suspected or confirmed sepsis
* Irregular heart rate, rhythm
* Receiving pressors to maintain blood pressure
* Presently implanted electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant
* Allergy to local anesthetics used for placement of the lead
* History of lung cancer, emphysema, chronic obstructive pulmonary disease, or other comorbidity that might otherwise compromise the expected air flow volumes in the lungs
* At risk of imminent respiratory collapse

  * Lung Function: FEV1 < 40% predicted
  * Signs and Symptoms: Extreme symptoms at rest, accessory muscle use, chest retraction
  * Alert State: Drowsy, confused
* Treatment with anti-cholinergic medications within 4 hours of enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JP Errico, Study Director — ElectroCore INC
Locations (6):
- United States (6):
  - Rush University Medical Center, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, Barnes-Jewish Hospital,, St Louis, Missouri
  - Dorrington Medical Associates, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resolve Stimulator and Proximity Lead
Started | 25
Completed | 23
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Safety population
Arm/Group | Resolve Stimulator and Proximity Lead
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 41 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 18
  Hispanic and white | 1
  American Indian or Alaska Native | 1
  White | 2
  Other | 1
  Hispanic Latino | 1
  Hispanic Black | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Safety- Number of Participants With Adverse Events
Description: Safety- Number of participants that reported Adverse Events
Time Frame: 2 weeks
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Resolve Stimulator and Proximity Lead
Number analyzed (Participants) | 25
Participants | 16

2. Secondary Outcome: Improvement of Common Measures of Breathing Performance, Forced Expiry Volume in 1second (FEV1).
Description: An assessment of Forced Expiry Volume in 1second (FEV1) measurements were taken throughout the course of treatment (15,30 and 60 minutes).
  Peak FEV1 measurements were recorded for each subject, and the number of minutes the subject had received treatment at the time of peak FEV1.
  The threshold for improvement was set at 12% over baseline at any of the time points (15,30 and 60 minutes). Outcome measure data indicates the number of subjects above 12%.
Time Frame: 60 minutes
Population: Safety population. 1 subject result missing due to no stimulation performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Resolve Stimulator and Proximity Lead
Number analyzed (Participants) | 24
Participants | 19

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Resolve Stimulator and Proximity Lead
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 11/25
Other Adverse Events (participants affected / at risk) | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resolve Stimulator and Proximity Lead (N=25)
Hospitalization for chest pain associated with cocaine use (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hospitalization for persistant asthma symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Death at 15 days post treatment (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for observation; respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for continuation of asthma exacerbation (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resolve Stimulator and Proximity Lead (N=25)
Muscle twitching in neck (Musculoskeletal and connective tissue disorders) | 3 (4)
Sweating during attempted lead advancement (Endocrine disorders) | 1 (1)
Lead displacement (Surgical and medical procedures) | 1 (1)
Neck pain for 2 days post treatment (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Bleeding at insertion site (Vascular disorders) | 1 (1)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less